CLINICAL TRIAL: NCT01656759
Title: Use of a Novel Fibrin Sealant in Total Knee Arthroplasty: A Prospective Randomized Controlled Clinical Trial
Brief Title: Use of a Novel Fibrin Sealant in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brett Levine, MD, Assistant Professor and Associate Residency Director, Rush University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 12032202-IRB01
Record Dates: First submitted 2012-06-14; First posted 2012-08-03 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis; Intraoperative Bleeding
Keywords: Blood Loss; Hemoglobin; Hematocrit; Blood Transfusions
MeSH Terms: conditions — Osteoarthritis; Blood Loss, Surgical; Hemorrhage | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Control group. Will not receive the fibrin spray.
- Treatment Group--Evicel Fibrin Spray (Active Comparator): Patient will receive the fibrin spray after implantation of device but before the wound is closed.
  Patients will be randomized to receive spray or not and postop parameters measured.
  Interventions: Drug: Evicel Fibrin Spray

INTERVENTIONS:
Drug: Evicel Fibrin Spray — 10cc syringe dose, once at the end of TKA
  Other Names: Produced by OMRIX Biopharmaceuticals, Ltd.
  Arms: Treatment Group--Evicel Fibrin Spray

SUMMARY:
Applying a fibrin spray, after knee device implantation, will help in reducing patient blood loss and decrease the drop in both hemoglobin and hematocrit levels. Also, with decreased blood loss there should be a reduced need for blood transfusions.

DETAILED DESCRIPTION:
Study Design

Study design and control methods:

This study is designed as a prospective, randomized, double-blinded controlled clinical trial to compare the effect of a fibrin spray applied to the surgical wound as compared to patients not receiving the fibrin spray.

Treatment group:

The subjects will be randomly assigned to the fibrin treatment group or to the control group at the time of the surgery via the opening of a randomly selected sealed envelope. The patient and the independent reviewer will be blinded as to which treatment group the patient is assigned to. This information will be linked to a confidential database for later review by the principal investigator.

Treatment allocation:

All eligible patients (i.e., meeting inclusion criteria and no exclusion criteria) will be treated and observed per the research protocol. All patients will maintain the right to refuse participation and receive a specific treatment of the study if desired.

Trial Population:

The target sample size is 70 patients for both the treatment and control groups (140 total) with each group split evenly between males and females. There will be one actively enrolling surgeon (Dr. Brett Levine). The goal is to enroll a total of 140 subjects experiencing joint pain that warrants a Total knee arthroplasty (TKA). The specific diagnosis for the joint pain will not direct the subjects' assignment or eligibility at the time of surgery. All 140 patients will be enrolled from the office of the primary investigator (Dr. Brett Levine). All indications for TKA will be included unless one of the exclusion criteria is met.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female of any race
* Ages 18-80 years old
* Patients must be undergoing an elective, primary knee arthroplasty performed by the principal investigator

Exclusion Criteria:

* Allergy or intolerance to the study materials
* Surgical intervention during the past month for the treatment of the painful joint or its underlying etiology
* History of previous surgeries on the affected joint including previous arthroscopy (open surgeries)
* Women that are pregnant or may become pregnant
* Patient declines to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett R Levine, MD, Principal Investigator — RUMC
Locations (1):
- Rush Oak Park Hospital, Oak Park, Illinois, United States

REFERENCES:
- [Result] Levy O, Martinowitz U, Oran A, Tauber C, Horoszowski H. The use of fibrin tissue adhesive to reduce blood loss and the need for blood transfusion after total knee arthroplasty. A prospective, randomized, multicenter study. J Bone Joint Surg Am. 1999 Nov;81(11):1580-8. doi: 10.2106/00004623-199911000-00010. PMID 10565650
- [Result] Wang GJ, Hungerford DS, Savory CG, Rosenberg AG, Mont MA, Burks SG, Mayers SL, Spotnitz WD. Use of fibrin sealant to reduce bloody drainage and hemoglobin loss after total knee arthroplasty: a brief note on a randomized prospective trial. J Bone Joint Surg Am. 2001 Oct;83(10):1503-5. doi: 10.2106/00004623-200110000-00007. PMID 11679600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, 21 patients were disqualified for protocol violation.
Groups:
- Treatment Group--Evicel Fibrin Spray: Patient will receive the fibrin spray after implantation of device but before the wound is closed.
  Patients will be randomized to receive spray or not and postop parameters measured.
  Evicel Fibrin Spray: 10cc syringe dose, once at the end of TKA
Period: Overall Study
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Started | 27 | 25
Completed | 25 | 22
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 64 (10) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Primary--Percent Change of Pre- to Post-Operative Hemoglobin
Description: Pre-operative hemoglobin values from routine CBC no earlier than 1 month prior to surgery were compared to post-operative hemoglobin values from routine CBC after surgery.
Time Frame: Pre-operative to 1 month
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Number analyzed (Participants) | 25 | 22
Percent Change | 20.1 (7.0) | 22.5 (5.7)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group--Evicel Fibrin Spray; Test type: Superiority or Other; p = 0.2, t-test, 2 sided

2. Primary Outcome: Total Blood Loss
Description: Combination of intraoperative and postoperative blood loss for participants.
Time Frame: Collected during surgery and in first 2-3 days after surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Number analyzed (Participants) | 25 | 22
mL | 605 (288) | 621 (334)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group--Evicel Fibrin Spray; Test type: Superiority or Other; p = 0.9, t-test, 2 sided

3. Secondary Outcome: Total Transfusions
Description: The number of transfusions each patient receives during their postoperative hospitalization.
Time Frame: 3 days
Measure: Number; unit: Number of transfusions
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Number analyzed (Participants) | 25 | 22
Number of transfusions | 3 | 3

4. Secondary Outcome: Postoperative Blood Loss
Description: Measured as drainage output from postoperative drains during hospitalization.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Number analyzed (Participants) | 25 | 22
mL | 543 (273) | 555 (324)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group--Evicel Fibrin Spray; Test type: Superiority or Other; p = 0.9, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Control Group | Treatment Group--Evicel Fibrin Spray
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=27) | Treatment Group--Evicel Fibrin Spray (N=25)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=27) | Treatment Group--Evicel Fibrin Spray (N=25)
Superficial Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes